CLINICAL TRIAL: NCT06554444
Title: Assessment of Volumetric Changes During the Early Healing Period of Dental Implant Treatment: Clinical, Radiographic, and Digital Evaluation
Brief Title: Assessment of Early Healing Period of Dental Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Assistant Professor, Kutahya Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 05
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant; Osseointegration; Biological Width

STUDY DESIGN:
Intervention Model Description: Dental implant placement in the posterior mandible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental implant placement in the posterior mandible (Experimental): In this study, patients who have tooth loss in the posterior mandible and meet the inclusion criteria will receive dental implants under local anesthesia
  Interventions: Procedure: Dental Implant Surgery

INTERVENTIONS:
Procedure: Dental Implant Surgery — Dental implants will be placed in edentulous areas.

SUMMARY:
This prospective cohort study aimed to evaluate, clinically, radiographically, and digitally, the volumetric changes occurring during the early healing period after implant treatment in patients with tooth loss in the posterior regions of the jaws, focusing on the processes of osseointegration and biological width formation.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Systemically healthy
* Need for implant treatment in unilaterally edentulous posterior mandible
* Sufficient interocclusal space for implant and restoration placement
* At least four months passed since tooth extraction
* Alveolar bone height adequate for implant placement, with a minimum width of 6 mm, and without risking anatomical structures
* Plaque and bleeding scores of less than 15% in the entire mouth
* Presence of opposing teeth in occlusion
* Written informed consent obtained, including permission for the use of data for research purposes

Exclusion Criteria:

* Poor oral hygiene
* Uncontrolled periodontal disease
* Pregnancy or lactation at any stage of the study
* Uncontrolled diabetes
* Patients with suppressed immune systems
* History of radiotherapy to the head and neck region
* Diseases or medications affecting bone metabolism
* Smoking more than 10 cigarettes per day
* Bone augmentation performed before or concurrently with the implant
* Failure to achieve primary stability with the implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Linear and volumetric changes in the tissue | Preoperative and postoperative 2nd, 4th, and 16th months
  Linear and volumetric changes in the tissue resulting from the alignment of scan data obtained at four different time points.

SECONDARY OUTCOMES:
Keratinized mucosa width (from the edentulous ridge) | Preoperative and postoperative 2nd month
  Keratinized tissue measured from the mid-buccal of the edentulous area using a periodontal probe.
Keratinized mucosa width (from the gingival margin of the dental implant-supported prosthesis) | Postoperative 4th and 16th months
  Keratinized tissue measured from the gingival margin of the dental implant-supported prosthesis to the mucogingival junction using a periodontal probe.
Mucosal thickness (from the edentulous ridge) | Preoperative and postoperative 2nd month
  Mucosal thickness measured from the midpoint of the edentulous area using a periodontal probe.
Mucosal thickness (from the facial aspect of the edentulous ridge) | Preoperative and postoperative 2nd month
  Mucosal thickness measured at the mid-buccal of the edentulous area, from the midpoint between the mucogingival junction and 2 mm apical to the gingival margin of the adjacent tooth, using a endodontic spreader.
Mucosal thickness (from 3 mm apical to the gingival margin of the implant-supported prosthesis) | Postoperative 4th and 16th months
  Mucosal thickness measured 3 mm apical to the gingival margin of the implant-supported prosthesis using a endodontic spreader.
Peri-implant pocket depth | Postoperative 4th and 16th months
  Peri-implant pocket depth measured at six points around the dental implant using a periodontal probe.
Modified plaque index | Postoperative 4th and 16th months
  Modified plaque index measured at four points around the dental implant using a periodontal probe.
Modified bleeding index | Postoperative 4th and 16th months
  Modified bleeding index measured at four points around the dental implant using a periodontal probe.
Marginal bone level | Preoperative and postoperative 2nd, 4th, and 16th months
  Marginal bone level measured on periapical radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tavelli L, Barootchi S, Vera Rodriguez M, Mancini L, Meneghetti PC, Mendonca G, Wang HL. Early soft tissue changes following implant placement with or without soft tissue augmentation using a xenogeneic cross-link collagen scaffold: A volumetric comparative study. J Esthet Restor Dent. 2022 Jan;34(1):181-187. doi: 10.1111/jerd.12856. Epub 2021 Dec 22. PMID 34936177